CLINICAL TRIAL: NCT05553041
Title: Evaluation of 18F-Fluciclovine PET-MRI to Differentiate Tumor Progression From Post-treatment Changes in Pediatric High-grade Glioma (HGG)
Brief Title: 18F-Fluciclovine PET-MRI in High-grade Glioma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Blue Earth Diagnostics (Industry); Dragon Master Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-019514
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Glioma; High Grade Glioma; Glioma, Malignant; Glioma Intracranial; Diffuse Glioma
Keywords: Glioma; High Grade Glioma; Glioma, Malignant; Glioma Intracranial; Diffuse Glioma; 18F fluciclovine
MeSH Terms: conditions — Glioma | interventions — fluciclovine F-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-Fluciclovine PET-MRI in pediatric HGG or DMG participants (Experimental): Single intravenous administration of 18F fluciclovine for PET-MRI Scan
  Interventions: Drug: 18F-Fluciclovine PET-MRI

INTERVENTIONS:
Drug: 18F-Fluciclovine PET-MRI — 18F-Fluciclovine will be injected via IV prior to Positron emission tomography (PET)-Magnetic resonance imaging (MRI)
  Other Names: Axumin

SUMMARY:
The purpose of this study is to see if 18F-fluciclovine (Axumin®) PET imaging is useful and safe in the management of children with High Grade Gliomas. Investigators seek to determine if this imaging will help doctors tell the difference between tumor growth (progression) and other tumor changes that can occur after treatment.

DETAILED DESCRIPTION:
Following radiation and immunotherapy, many pediatric participants with high-grade gliomas (HGG), including diffuse midline glioma (DMG), demonstrate radiographic findings suspicious of disease progression. Differentiating post-treatment changes from true tumor progression is paramount to clinical decision-making, as true tumor progression may warrant a change in treatment, while post-treatment changes are typically not an indication to change treatment. Unfortunately, conventional MRI cannot reliably distinguish between true progression and post-treatment changes. Therefore, finding a physiological correlate to delineate true progression from pseudo-progression is critical.

The overall objective of this current application is to evaluate 18F-fluciclovine PET imaging as a diagnostic biomarker for tumor progression compared to post-treatment changes in pediatric HGG. The long-term goal of this research is to accurately differentiate tumor progression from post-treatment changes in pediatric HGG using 18F-fluciclovine PET imaging.

ELIGIBILITY:
Inclusion Criteria

* 1. Histopathology-proven HGG (WHO grade III-IV) or DMG (WHO grade IV) or, in the case of DMG of the pons, imaging that is characteristic of Diffuse intrinsic pontine gliomas (DIPG) (diffusely infiltrating >=2/3 of the pons).
* 2. Measurable disease, measuring at least 1x1 cm.
* 3. Life expectancy of greater than 8 weeks.
* 4. Age > 1 years but < 21 years of age at enrollment.

For those without planned surgery:

* 1. Participants with clinical and/or radiographic suspicion of True progression (TP) or Pseudoprogression (PsP) during radiation but yet to have the initial post-radiation MRI scan.

or

* 2. Participants with suspicion for TP or PsP on first post-radiation MRI

For those with planned surgery:

* 1. Clinical or radiographic suspicion of tumor progression with plan to undergo surgery or biopsy.

Exclusion Criteria:

* 1. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician.
* 2. Pregnant or breastfeeding participants.
* 3. Participant who would require sedation or anesthesia for imaging beyond standard of care (SOC).
* 4. Participants who weigh less than 8 kg.
* 5. Participants who cannot avoid contact with a pregnant woman or infant for at least 12 hours following injection.
* 6. Participants with a history of abnormal kidney function or creatinine >= CTCAE v5.0 grade 2 at time of study registration.

  7. Participants with primary tumors of the spinal cord.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Image analysis | 6 months
  Comparison of Standardized uptake value (SUV) max, SUV peak, and uptake kinetics post radiation between participants who experience true progression versus those who experience pseudoprogression as confirmed by routine imaging.
Histopathology analysis | 4 weeks
  Evaluation of SUV uptake post radiation in participants with planned biopsy or resection who experience true progression versus those who experience pseudoprogression as confirmed by histopathology.

SECONDARY OUTCOMES:
Safety of 18F-Fluciclovine | 6 months
  The Safety profile of 18F-Fluciclovine PET in pediatric HGG participants will be assessed based on CTCAE 5.0 toxicity experienced after administration of 18F-Fluciclovine

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Aboian, MD,PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calmon R, Puget S, Varlet P, Dangouloff-Ros V, Blauwblomme T, Beccaria K, Grevent D, Sainte-Rose C, Castel D, Debily MA, Dufour C, Bolle S, Dhermain F, Saitovitch A, Zilbovicius M, Brunelle F, Grill J, Boddaert N. Cerebral blood flow changes after radiation therapy identifies pseudoprogression in diffuse intrinsic pontine gliomas. Neuro Oncol. 2018 Jun 18;20(7):994-1002. doi: 10.1093/neuonc/nox227. PMID 29244086
- [Background] Carceller F, Fowkes LA, Khabra K, Moreno L, Saran F, Burford A, Mackay A, Jones DT, Hovestadt V, Marshall LV, Vaidya S, Mandeville H, Jerome N, Bridges LR, Laxton R, Al-Sarraj S, Pfister SM, Leach MO, Pearson AD, Jones C, Koh DM, Zacharoulis S. Pseudoprogression in children, adolescents and young adults with non-brainstem high grade glioma and diffuse intrinsic pontine glioma. J Neurooncol. 2016 Aug;129(1):109-21. doi: 10.1007/s11060-016-2151-8. Epub 2016 May 14. PMID 27180091
- [Background] Vajapeyam S, Brown D, Billups C, Patay Z, Vezina G, Shiroishi MS, Law M, Baxter P, Onar-Thomas A, Fangusaro JR, Dunkel IJ, Poussaint TY. Advanced ADC Histogram, Perfusion, and Permeability Metrics Show an Association with Survival and Pseudoprogression in Newly Diagnosed Diffuse Intrinsic Pontine Glioma: A Report from the Pediatric Brain Tumor Consortium. AJNR Am J Neuroradiol. 2020 Apr;41(4):718-724. doi: 10.3174/ajnr.A6499. Epub 2020 Apr 2. PMID 32241771
- [Background] Bhutia YD, Babu E, Ramachandran S, Ganapathy V. Amino Acid transporters in cancer and their relevance to "glutamine addiction": novel targets for the design of a new class of anticancer drugs. Cancer Res. 2015 May 1;75(9):1782-8. doi: 10.1158/0008-5472.CAN-14-3745. Epub 2015 Apr 8. PMID 25855379
- [Background] Galldiks N, Law I, Pope WB, Arbizu J, Langen KJ. The use of amino acid PET and conventional MRI for monitoring of brain tumor therapy. Neuroimage Clin. 2016 Dec 18;13:386-394. doi: 10.1016/j.nicl.2016.12.020. eCollection 2017. PMID 28116231
- [Background] Oka S, Hattori R, Kurosaki F, Toyama M, Williams LA, Yu W, Votaw JR, Yoshida Y, Goodman MM, Ito O. A preliminary study of anti-1-amino-3-18F-fluorocyclobutyl-1-carboxylic acid for the detection of prostate cancer. J Nucl Med. 2007 Jan;48(1):46-55. PMID 17204698
- [Background] Oka S, Okudaira H, Ono M, Schuster DM, Goodman MM, Kawai K, Shirakami Y. Differences in transport mechanisms of trans-1-amino-3-[18F]fluorocyclobutanecarboxylic acid in inflammation, prostate cancer, and glioma cells: comparison with L-[methyl-11C]methionine and 2-deoxy-2-[18F]fluoro-D-glucose. Mol Imaging Biol. 2014 Jun;16(3):322-9. doi: 10.1007/s11307-013-0693-0. PMID 24136390
- [Background] Zinnhardt B, Pigeon H, Theze B, Viel T, Wachsmuth L, Fricke IB, Schelhaas S, Honold L, Schwegmann K, Wagner S, Faust A, Faber C, Kuhlmann MT, Hermann S, Schafers M, Winkeler A, Jacobs AH. Combined PET Imaging of the Inflammatory Tumor Microenvironment Identifies Margins of Unique Radiotracer Uptake. Cancer Res. 2017 Apr 15;77(8):1831-1841. doi: 10.1158/0008-5472.CAN-16-2628. Epub 2017 Jan 30. PMID 28137769
- [Background] Henderson F Jr, Brem S, O'Rourke DM, Nasrallah M, Buch VP, Young AJ, Doot RK, Pantel A, Desai A, Bagley SJ, Nabavizadeh SA. 18F-Fluciclovine PET to distinguish treatment-related effects from disease progression in recurrent glioblastoma: PET fusion with MRI guides neurosurgical sampling. Neurooncol Pract. 2020 Mar;7(2):152-157. doi: 10.1093/nop/npz068. Epub 2019 Dec 8. PMID 32206320
- [Background] Galldiks N, Dunkl V, Stoffels G, Hutterer M, Rapp M, Sabel M, Reifenberger G, Kebir S, Dorn F, Blau T, Herrlinger U, Hau P, Ruge MI, Kocher M, Goldbrunner R, Fink GR, Drzezga A, Schmidt M, Langen KJ. Diagnosis of pseudoprogression in patients with glioblastoma using O-(2-[18F]fluoroethyl)-L-tyrosine PET. Eur J Nucl Med Mol Imaging. 2015 Apr;42(5):685-95. doi: 10.1007/s00259-014-2959-4. Epub 2014 Nov 20. PMID 25411133
- [Background] Nihashi T, Dahabreh IJ, Terasawa T. Diagnostic accuracy of PET for recurrent glioma diagnosis: a meta-analysis. AJNR Am J Neuroradiol. 2013 May;34(5):944-50, S1-11. doi: 10.3174/ajnr.A3324. Epub 2012 Nov 1. PMID 23124638
- [Background] Songmen S, Nepal P, Olsavsky T, Sapire J. Axumin Positron Emission Tomography: Novel Agent for Prostate Cancer Biochemical Recurrence. J Clin Imaging Sci. 2019 Nov 6;9:49. doi: 10.25259/JCIS_139_2019. eCollection 2019. PMID 31819826
- [Background] Wakabayashi T, Iuchi T, Tsuyuguchi N, Nishikawa R, Arakawa Y, Sasayama T, Miyake K, Nariai T, Narita Y, Hashimoto N, Okuda O, Matsuda H, Kubota K, Ito K, Nakazato Y, Kubomura K. Diagnostic Performance and Safety of Positron Emission Tomography Using 18F-Fluciclovine in Patients with Clinically Suspected High- or Low-grade Gliomas: A Multicenter Phase IIb Trial. Asia Ocean J Nucl Med Biol. 2017 Winter;5(1):10-21. doi: 10.22038/aojnmb.2016.7869. PMID 28840134
- [Background] Shoup TM, Olson J, Hoffman JM, Votaw J, Eshima D, Eshima L, Camp VM, Stabin M, Votaw D, Goodman MM. Synthesis and evaluation of [18F]1-amino-3-fluorocyclobutane-1-carboxylic acid to image brain tumors. J Nucl Med. 1999 Feb;40(2):331-8. PMID 10025843
- [Background] Michaud L, Beattie BJ, Akhurst T, Dunphy M, Zanzonico P, Finn R, Mauguen A, Schoder H, Weber WA, Lassman AB, Blasberg R. 18F-Fluciclovine (18F-FACBC) PET imaging of recurrent brain tumors. Eur J Nucl Med Mol Imaging. 2020 Jun;47(6):1353-1367. doi: 10.1007/s00259-019-04433-1. Epub 2019 Aug 15. PMID 31418054
- [Background] Tsuyuguchi N, Terakawa Y, Uda T, Nakajo K, Kanemura Y. Diagnosis of Brain Tumors Using Amino Acid Transport PET Imaging with 18F-fluciclovine: A Comparative Study with L-methyl-11C-methionine PET Imaging. Asia Ocean J Nucl Med Biol. 2017 Spring;5(2):85-94. doi: 10.22038/aojnmb.2017.8843. PMID 28660218
- [Background] Parent EE, Benayoun M, Ibeanu I, Olson JJ, Hadjipanayis CG, Brat DJ, Adhikarla V, Nye J, Schuster DM, Goodman MM. [18F]Fluciclovine PET discrimination between high- and low-grade gliomas. EJNMMI Res. 2018 Jul 25;8(1):67. doi: 10.1186/s13550-018-0415-3. PMID 30046944
- [Background] Kondo A, Ishii H, Aoki S, Suzuki M, Nagasawa H, Kubota K, Minamimoto R, Arakawa A, Tominaga M, Arai H. Phase IIa clinical study of [18F]fluciclovine: efficacy and safety of a new PET tracer for brain tumors. Ann Nucl Med. 2016 Nov;30(9):608-618. doi: 10.1007/s12149-016-1102-y. Epub 2016 Jul 14. PMID 27418267
- [Background] Liu CJ, Lu MY, Liu YL, Ko CL, Ko KY, Tzen KY, Chang HH, Yang YL, Jou ST, Hsu WM, Yen RF. Risk Stratification of Pediatric Patients With Neuroblastoma Using Volumetric Parameters of 18F-FDG and 18F-DOPA PET/CT. Clin Nucl Med. 2017 Mar;42(3):e142-e148. doi: 10.1097/RLU.0000000000001529. PMID 28072621
- [Background] Marner L, Nysom K, Sehested A, Borgwardt L, Mathiasen R, Henriksen OM, Lundemann M, Munck Af Rosenschold P, Thomsen C, Bogeskov L, Skjoth-Rasmussen J, Juhler M, Kruse A, Broholm H, Scheie D, Lauritsen T, Forman JL, Wehner PS, Hojgaard L, Law I. Early Postoperative 18F-FET PET/MRI for Pediatric Brain and Spinal Cord Tumors. J Nucl Med. 2019 Aug;60(8):1053-1058. doi: 10.2967/jnumed.118.220293. Epub 2019 Jan 25. PMID 30683767
- [Background] Morana G, Piccardo A, Puntoni M, Nozza P, Cama A, Raso A, Mascelli S, Massollo M, Milanaccio C, Garre ML, Rossi A. Diagnostic and prognostic value of 18F-DOPA PET and 1H-MR spectroscopy in pediatric supratentorial infiltrative gliomas: a comparative study. Neuro Oncol. 2015 Dec;17(12):1637-47. doi: 10.1093/neuonc/nov099. Epub 2015 Sep 23. PMID 26405202
- [Background] Albert NL, Weller M, Suchorska B, Galldiks N, Soffietti R, Kim MM, la Fougere C, Pope W, Law I, Arbizu J, Chamberlain MC, Vogelbaum M, Ellingson BM, Tonn JC. Response Assessment in Neuro-Oncology working group and European Association for Neuro-Oncology recommendations for the clinical use of PET imaging in gliomas. Neuro Oncol. 2016 Sep;18(9):1199-208. doi: 10.1093/neuonc/now058. Epub 2016 Apr 21. PMID 27106405
- [Background] Werner JM, Lohmann P, Fink GR, Langen KJ, Galldiks N. Current Landscape and Emerging Fields of PET Imaging in Patients with Brain Tumors. Molecules. 2020 Mar 24;25(6):1471. doi: 10.3390/molecules25061471. PMID 32213992
- [Background] Law I, Albert NL, Arbizu J, Boellaard R, Drzezga A, Galldiks N, la Fougere C, Langen KJ, Lopci E, Lowe V, McConathy J, Quick HH, Sattler B, Schuster DM, Tonn JC, Weller M. Joint EANM/EANO/RANO practice guidelines/SNMMI procedure standards for imaging of gliomas using PET with radiolabelled amino acids and [18F]FDG: version 1.0. Eur J Nucl Med Mol Imaging. 2019 Mar;46(3):540-557. doi: 10.1007/s00259-018-4207-9. Epub 2018 Dec 5. PMID 30519867
- [Background] Bashir A, Mathilde Jacobsen S, Molby Henriksen O, Broholm H, Urup T, Grunnet K, Andree Larsen V, Moller S, Skjoth-Rasmussen J, Skovgaard Poulsen H, Law I. Recurrent glioblastoma versus late posttreatment changes: diagnostic accuracy of O-(2-[18F]fluoroethyl)-L-tyrosine positron emission tomography (18F-FET PET). Neuro Oncol. 2019 Dec 17;21(12):1595-1606. doi: 10.1093/neuonc/noz166. PMID 31618420
- [Background] Galldiks N, Stoffels G, Filss C, Rapp M, Blau T, Tscherpel C, Ceccon G, Dunkl V, Weinzierl M, Stoffel M, Sabel M, Fink GR, Shah NJ, Langen KJ. The use of dynamic O-(2-18F-fluoroethyl)-l-tyrosine PET in the diagnosis of patients with progressive and recurrent glioma. Neuro Oncol. 2015 Sep;17(9):1293-300. doi: 10.1093/neuonc/nov088. Epub 2015 May 24. PMID 26008606
- [Background] Herrmann K, Czernin J, Cloughesy T, Lai A, Pomykala KL, Benz MR, Buck AK, Phelps ME, Chen W. Comparison of visual and semiquantitative analysis of 18F-FDOPA-PET/CT for recurrence detection in glioblastoma patients. Neuro Oncol. 2014 Apr;16(4):603-9. doi: 10.1093/neuonc/not166. Epub 2013 Dec 4. PMID 24305722
- [Background] Kebir S, Fimmers R, Galldiks N, Schafer N, Mack F, Schaub C, Stuplich M, Niessen M, Tzaridis T, Simon M, Stoffels G, Langen KJ, Scheffler B, Glas M, Herrlinger U. Late Pseudoprogression in Glioblastoma: Diagnostic Value of Dynamic O-(2-[18F]fluoroethyl)-L-Tyrosine PET. Clin Cancer Res. 2016 May 1;22(9):2190-6. doi: 10.1158/1078-0432.CCR-15-1334. Epub 2015 Dec 16. PMID 26673798